CLINICAL TRIAL: NCT01436591
Title: Comparison of Diagnostic Performance of an Algorithm and a High Definition Classical Iterative Algorithm Positron Emission Tomography (PET) to 18Fluoro-deoxy-glucose (18FDG) in the Evaluation of Axillary Lymph Node Invasion of Breast Tumors
Acronym: TEP-Sein
Status: Terminated | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: TEP-Sein
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast; 18FDG; Axillary; Positron Emission Tomography
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary endpoint of this study is to show that this algorithm in high definition is superior to the classical algorithm in the diagnosis of lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and signed by the patient
* Age ≥ 18 years
* Breast tumor for which the therapeutic indication for surgery has from the outset: breast surgery (conservative or radical) associated with a conventional axillary dissection
* Proof of infiltrating ductal carcinoma histology
* No known metastasis
* No cons-indication to anesthesia.

Exclusion criteria:

* History of neoadjuvant therapy
* Patients with invasive lobular carcinoma
* Indication of the use of sentinel node (if invasive carcinoma uni-centric, ≤ 2 cm in diameter, without palpable lymphadenopathy (N0))
* Diabetes is not controlled by conventional treatment (blood glucose> 1.8 g / l)
* Inability to capital
* Patients who are pregnant or nursing or of childbearing potential and not using adequate contraception
* Persons deprived of their liberty
* Major subject of a measure of legal protection or unable to consent
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preoperative assessment of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Performance of FDG-PET for the evaluation of nodal status | 3 years
  Show that the algorithm of high-definition positron emission tomography (PET) to 18Fluoro-deoxy-glucose (18FDG) is greater than a classical algorithm in the diagnosis of lymph node metastases.

SECONDARY OUTCOMES:
Information on lymph node status in patients with breast cancer. | 3 years
  Show that scintigraphy performed on a FDG positron camera equipped with a reconstruction algorithm for high-definition can provide reliable information on lymph node status in patients with breast cancer and determine the minimum size of lymph node metastatic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: SWITSERS Odile, Dr, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François Baclesse, Caen, France